CLINICAL TRIAL: NCT01308801
Title: Benefice Assessment of Repetitive Transcranial Magnetic Stimulation Used as an Additional Procedure to Rehabilitation Exercises in Patients Suffering From Fibromyalgia
Brief Title: Repetitive Transcranial Magnetic Stimulation in Fibromyalgia
Acronym: STIMALGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-A00865-34
Record Dates: First submitted 2010-12-17; First posted 2011-03-04 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2016-01

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pain; repetitive transcranial magnetic stimulation; rehabilitation exercise; quality of life
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active rTMS + rehabilitation exercise (Experimental): 14 weeks of active repetitive transcranial magnetic stimulation associated with rehabilitation exercise
  Interventions: Device: active rTMS + rehabilitation exercise
- placebo rTMS + rehabilitation exercise (Placebo Comparator): 14 weeks of placebo repetitive transcranial magnetic stimulation associated with rehabilitation exercise
  Interventions: Device: placebo rTMS+ rehabilitation exercise

INTERVENTIONS:
Device: active rTMS + rehabilitation exercise — 14 weeks program of active repetitive transcranial magnetic stimulation associated with rehabilitation exercise
  Arms: active rTMS + rehabilitation exercise
Device: placebo rTMS+ rehabilitation exercise — 14 week program of placebo repetitive transcranial magnetic stimulation associated with rehabilitation exercise
  Arms: placebo rTMS + rehabilitation exercise

SUMMARY:
The purpose of this study is to determine the analgesic effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) used as an additional procedure to rehabilitation exercises in patient suffering from fibromyalgia.

A double blind clinical trial with two randomized parallel groups:

* Placebo rTMS and rehabilitation exercise
* Active rTMS and rehabilitation exercise

DETAILED DESCRIPTION:
Fibromyalgia is the most frequent chronic diffuse painful disease (3 to 4% of the general population).

Analgesic drugs are widely used in fibromyalgia, pain being the main symptom. However the effectiveness of analgesic drugs is often insufficient.

Among non-drug therapies, rehabilitation exercise plays an important role with a special interest in terms of the quality of life, strain and pain.

More recently the Transcranial Magnetic Stimulation effects have been evaluated in patients suffering from fibromyalgia with a statistically significative analgesic effect.

Both rehabilitation exercise and Transcranial Magnetic Stimulation (rTMS) have shown their respective analgesic effectiveness in fibromyalgia. It now seems important to evaluate the combination of these two therapies.

Main objective: To evaluate the analgesic effect of rTMS in fibromyalgia patients doing rehabilitation exercise.

Primary endpoint:

The evaluation methode used is a visual analog scale (VAS) of pain. Patients will note down every day VAS of over the last 24 hours.

The evolution of the VAS during the treatment period with respect to baseline, will be compared in both groups, active rTMS and placebo rTMS.

The investigators will analyze the average daily VAS for different weeks (W2, W4, W8, W14) compared to the average daily VAS at the baseline.

After a baseline period of 15 days, patients will begin sessions of rTMS and rehabilitation exercise for a period of 14 weeks.

The study is composed of three assessment visits : a baseline visit, a visit corresponding to the end of the therapy with exercise period and a last assessment visit at 26 weeks after the end of the treatment.

These visits will include clinical examination, blood test, an effort test, an orthostatic test, a resistance to fatigue test and polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* primary fibromyalgia according to the American College of Rheumatology
* no contraindication to rehabilitation exercise
* pain with VAS > 4 during at least six months
* FIQ score > 50
* no change in drug therapy over the last month
* affiliation to French Health Service

Exclusion Criteria:

* BMI > 35kg/m²
* patient who has already benefited from rTMS
* rTMS contraindication
* restless legs symptom
* patient suffering from major depression
* patient suffering from inflammatory rheumatism, autoimmune disease, other chronic pain pathology
* sleep apnea syndrome
* no contraindication to rTMS or MRI
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain Visual Analog Scale (VAS) at 14 weeks of treatment | Daily average VAS at baseline, week 2, week 4, week 8, week 14
  Patient will note down each day the VAS for the last 24 hours.

SECONDARY OUTCOMES:
Change from base line in quality of life at 14 weeks and 26 weeks | At the beginning of the program, at the end (14 weeks), and 26 weeks after the end of the program
  Fibromyalgia Impact Questionnaire (FIQ)
Change from base line in depression assessment at 14 weeks and 26 weeks | at the beginning of the program, at the end (14 weeks), and 26 weeks after the end of the program
  Beck Depression Inventory (BDI)
Change from baseline in Covi's anxiety scale | at the beginning of the program, at the end (14 weeks), and 26 weeks after the end of the program
  Covi's anxiety scale
Change from baseline in sleep quality at 14 weeks abd 26 weeks | At the beginning of the program, at the end (14 weeks), and 26 weeks after the end of the program
  Number of times awaking at night
Change from baseline in neuromuscular fatigability at 14 weeks and 26 weeks | At the beginning of the program, at the end (14 weeks), and 26 weeks after the end of the program
  Maximal voluntary activation level
Change from baseline in cardiac variability at 14 weeks and 26 weeks | At the beginning of the program, at the end (14 weeks), and 26 weeks after the end of the program
  RMSSD values, power of spectral density HF, KF, LF/HF, alpha index (baroreflex sensitivity)
Evolution of the analgesic effect after the end of the program | Daily average VAS at the end (14 weeks) and 26 weeks after the end of the program
  Patient will note down each day the VAS for the last 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Maindet-Dominici, MD, Principal Investigator — Centre de la Douleur CHU de Grenoble
Locations (1):
- CHU de Grenoble, Grenoble, Isère, France

REFERENCES:
- [Background] Burckhardt CS, Clark SR, Bennett RM. Fibromyalgia and quality of life: a comparative analysis. J Rheumatol. 1993 Mar;20(3):475-9. PMID 8478854
- [Background] Busch AJ, Schachter CL, Overend TJ, Peloso PM, Barber KA. Exercise for fibromyalgia: a systematic review. J Rheumatol. 2008 Jun;35(6):1130-44. Epub 2008 May 1. PMID 18464301
- [Background] Busch AJ, Barber KA, Overend TJ, Peloso PM, Schachter CL. Exercise for treating fibromyalgia syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003786. doi: 10.1002/14651858.CD003786.pub2. PMID 17943797
- [Background] Cook DB, Nagelkirk PR, Poluri A, Mores J, Natelson BH. The influence of aerobic fitness and fibromyalgia on cardiorespiratory and perceptual responses to exercise in patients with chronic fatigue syndrome. Arthritis Rheum. 2006 Oct;54(10):3351-62. doi: 10.1002/art.22124. PMID 17009309
- [Background] Dauvilliers Y, Touchon J. [Sleep in fibromyalgia: review of clinical and polysomnographic data]. Neurophysiol Clin. 2001 Feb;31(1):18-33. doi: 10.1016/s0987-7053(00)00240-9. French. PMID 11281066
- [Background] Passard A, Attal N, Benadhira R, Brasseur L, Saba G, Sichere P, Perrot S, Januel D, Bouhassira D. Effects of unilateral repetitive transcranial magnetic stimulation of the motor cortex on chronic widespread pain in fibromyalgia. Brain. 2007 Oct;130(Pt 10):2661-70. doi: 10.1093/brain/awm189. Epub 2007 Sep 14. PMID 17872930
- [Result] Guinot M, Maindet C, Hodaj H, Hodaj E, Bachasson D, Baillieul S, Cracowski JL, Launois S. Effects of Repetitive Transcranial Magnetic Stimulation and Multicomponent Therapy in Patients With Fibromyalgia: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2021 Mar;73(3):449-458. doi: 10.1002/acr.24118. PMID 31785190